CLINICAL TRIAL: NCT03734952
Title: Prospective Randomized Controlled Trial of Postoperative Radiotherapy in Thoracic Esophageal Squamous Cell Carcinoma With Neoadjuvant Chemoradiotherapy
Brief Title: Postoperative Radiotherapy in Thoracic Esophageal Squamous Cell Carcinoma With Neoadjuvant Chemoradiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Benhua Xu, Director,Radiation Oncology, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FujianUnionH-ESSC
Record Dates: First submitted 2018-10-26; First posted 2018-11-08 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Radiation Oncology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Neoadjuvant Radiotherapy Program+Neoadjuvant chemotherapy Program+ Esophagectomy program+Postoperative radiotherapy program
  Interventions: Radiation: Neoadjuvant Radiotherapy Program:; Drug: Neoadjuvant chemotherapy Program; Procedure: Esophagectomy program:; Radiation: Postoperative radiotherapy program
- Group B (Other): Neoadjuvant Radiotherapy Program+Neoadjuvant chemotherapy Program+ Esophagectomy program
  Interventions: Radiation: Neoadjuvant Radiotherapy Program:; Drug: Neoadjuvant chemotherapy Program; Procedure: Esophagectomy program:

INTERVENTIONS:
Radiation: Neoadjuvant Radiotherapy Program: — Gross tumor volume (GTV) should include the primary tumor and involved regional lymph nodes as identified on pre-treatment diagnostic studies. Clinical target volume (CTV) is defined as the primary tumor plus 3cm expansion superiorly and inferiorly along the length of the esophagus and a 1cm radial expansion.The nodal CTV should be defined by a 0.5cm expansion from the nodal GTV.CTV should also include coverage the nodal region(s) in which the involved lymph node(s). A total dose of 45 Gy in 25 fractions is delivered 5 days per week on workdays with intensity modulated radiotherapy (IMRT).
Drug: Neoadjuvant chemotherapy Program — Chemotherapy is delivered concomitantly and composed of two cycles of Docetaxel 60mg per square meter of body-surface area and cisplatin 75mg per square meter of body-surface area every 21 days at the intervals of neoadjuvant radiotherapy.
Procedure: Esophagectomy program: — Patients receive esophagectomy in 4-6 weeks after neoadjuvant neoadjuvant chemotherapy
Radiation: Postoperative radiotherapy program — A total dose of 18 Gy in10 fractions is delivered 5 days per week on workdays with IMRT.
  Arms: Group A

SUMMARY:
The primary objective is to compare surgery with postoperative radiotherapy (PORT) versus surgery, in terms of the overall survival time (OS) in Stage II or III squamous cell esophageal carcinoma with neoadjuvant chemoradiotherapy(nCRT).

DETAILED DESCRIPTION:
Esophageal squamous cell carcinoma (ESCC) is a common type of esophageal carcinoma in China, which is characterized by rapid development and fatal prognosis in most patients. Neoadjuvant chemoradiotherapy (nCRT) has been explored for many years in western countries and Japan, and proved to get survival benefit, especially for locally advanced esophageal cancer. However, the recurrence is the major cause of treatment failure in patients with ESCC. Our hypothesis is that inadequate radiation dose leads to recurrence of ESCC with nCRT and PORT lower recurrence rate and improved OS. As is known, there are no any studies concentrating on PORT in ESCC with nCRT. Patients are randomly assigned to PORT (Group A) or without PORT (Group B) with a 1:1 allocation ratio. The primary outcome is OS assessed with a minimum follow-up of 60 months. Secondary outcomes are progression-free survival (PFS), recurrence-free survival (RFS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must not have received any prior anticancer therapy Histologically-confirmed squamous cell carcinoma of the esophagus;
2. Tumors of the esophagus are located in the thoracic cavity;
3. Pre-treatment stageⅡ-Ⅲ (AJCC/UICC 8th Edition)
4. Male or non pregnant female
5. Age is between 18 years and 65 years,
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 or Karnofsky performance status (KPS) of 70 or more;
7. Adequate bone marrow function (White Blood Cells ≥4x109 /L; Neutrophil ≥1.5×109 /L; Hemoglobin≥ 90 g/L; platelets≥100x109 /L);
8. Adequate liver function (Total bilirubin, Aspartate transaminase(AST) and Alanine transaminase (ALT) ≤2x Upper Level of Normal (ULN));
9. Adequate renal function (serum creatinine (SCr) ≤1.5 x ULN);
10. The patient has provided written informed consent and is able to understand and comply with the study.

Exclusion Criteria:

1. Patients with non-squamous cell carcinoma histology;
2. Patients with advanced inoperable or metastatic esophageal cancer;
3. Patients with another previous or current malignant disease；
4. Any patient with a significant medical condition which is thought unlikely to tolerate the therapies. Such as cardiac disease;
5. Age >65 years;
6. Pregnant or lactating female or people during the birth-period who refused to take contraceptives;
7. Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior;
8. Patients who refuse surgery after neoadjuvant chemotherapy;
9. Unsuitable to be enrolled in the trial in the opinion of the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | From enrollment to 5 years after the end of treatment
  The length of time from enrollment until the time of death

SECONDARY OUTCOMES:
disease free survival | From enrollment to 5 years after the end of treatment
  The length of time from enrollment until the time of progression of disease
local recurrence rate | From enrollment to 5 years after the end of treatment
  The percent of the patient with local recurrence
Side effects | From enrollment to 12 weeks after end of the treatment
  adverse events according to NCI CTCAE 4.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Benhua Xu, doctor, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Yen YC, Chang JH, Lin WC, Chiou JF, Chang YC, Chang CL, Hsu HL, Chow JM, Yuan KS, Wu ATH, Wu SY. Effectiveness of esophagectomy in patients with thoracic esophageal squamous cell carcinoma receiving definitive radiotherapy or concurrent chemoradiotherapy through intensity-modulated radiation therapy techniques. Cancer. 2017 Jun 1;123(11):2043-2053. doi: 10.1002/cncr.30565. Epub 2017 Feb 2. PMID 28152166
- [Background] Burmeister BH, Thomas JM, Burmeister EA, Walpole ET, Harvey JA, Thomson DB, Barbour AP, Gotley DC, Smithers BM. Is concurrent radiation therapy required in patients receiving preoperative chemotherapy for adenocarcinoma of the oesophagus? A randomised phase II trial. Eur J Cancer. 2011 Feb;47(3):354-60. doi: 10.1016/j.ejca.2010.09.009. PMID 21084184
- [Background] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Background] Cao XF, He XT, Ji L, Xiao J, Lv J. Effects of neoadjuvant radiochemotherapy on pathological staging and prognosis for locally advanced esophageal squamous cell carcinoma. Dis Esophagus. 2009;22(6):477-81. doi: 10.1111/j.1442-2050.2008.00910.x. PMID 19703071
- [Background] Chen Y, Hao D, Wu X, Xing W, Yang Y, He C, Wang W, Liu J, Wang J. Neoadjuvant versus adjuvant chemoradiation for stage II-III esophageal squamous cell carcinoma: a single institution experience. Dis Esophagus. 2017 Jul 1;30(7):1-7. doi: 10.1093/dote/dox016. PMID 28475725
- [Background] Stahl M, Walz MK, Riera-Knorrenschild J, Stuschke M, Sandermann A, Bitzer M, Wilke H, Budach W. Preoperative chemotherapy versus chemoradiotherapy in locally advanced adenocarcinomas of the oesophagogastric junction (POET): Long-term results of a controlled randomised trial. Eur J Cancer. 2017 Aug;81:183-190. doi: 10.1016/j.ejca.2017.04.027. PMID 28628843
- [Background] van Hagen P, Hulshof MC, van Lanschot JJ, Steyerberg EW, van Berge Henegouwen MI, Wijnhoven BP, Richel DJ, Nieuwenhuijzen GA, Hospers GA, Bonenkamp JJ, Cuesta MA, Blaisse RJ, Busch OR, ten Kate FJ, Creemers GJ, Punt CJ, Plukker JT, Verheul HM, Spillenaar Bilgen EJ, van Dekken H, van der Sangen MJ, Rozema T, Biermann K, Beukema JC, Piet AH, van Rij CM, Reinders JG, Tilanus HW, van der Gaast A; CROSS Group. Preoperative chemoradiotherapy for esophageal or junctional cancer. N Engl J Med. 2012 May 31;366(22):2074-84. doi: 10.1056/NEJMoa1112088. PMID 22646630